CLINICAL TRIAL: NCT01546480
Title: From Acute to Chronic Postoperative Pain in Patients for Elective Cholecystectomy. Immunological Tests
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Vejle Hospital (Other); Oberstinde Kirsten Jensa la Cours Foundation (Other)
Responsible Party: Principal Investigator, Morten Rune Eckhardt, Afdelingslæge, Odense University Hospital
Other Study IDs: ImmT; 119 (Other: hhh)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: Chronic postoperative pain; Postcholecystectomy pain; Inflammation; Interleukines
MeSH Terms: conditions — Pain; Pain, Postoperative; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Serum Plasma Cerebrospinal fluid Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pain patients: Patients with unexplained chronic abdominal pain 12 months after elective cholecystectomy
- Operated painfree Patients: Painfree patients 12 months after elective cholecystectomy
- Nonoperated painfree patients: Painfree patients with no previous abdominal operation

SUMMARY:
Chronic Pain after Cholecystectomy is a well known problem. One theory is that it is due to persisting inflammation.

The purpose of the study is to measure inflammatory factors in cerebrospinal fluid and blod at patients 12 months after the operation.

DNA-samples are collected to examine genetical factors, important for perception of pain, and the development of chronic pain.

ELIGIBILITY:
Group 1:

Inclusion Criteria:

* Unexplained abdominal pain 12 months after elective cholecystectomy

Exclusion Criteria:

* Immunosuppressive treatment (NSAID excepted)
* Anticoagulant treatment

Group 2:

Inclusion Criteria:

* No pain 12 months after elective cholecystectomy

Exclusion Criteria:

* Immunosuppressive treatment (NSAID excepted)
* Anticoagulant treatment

Group 3:

Inclusion Criteria:

* Elective operation in spinal anesthesia or
* Or healthy volunteers accepting samples of blod, cerebral spinal fluid and saliva, to be collected

Exclusion Criteria:

* Acute or chronic pain condition
* Immunosuppressive treatment (NSAID excepted)
* Previous abdominal operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in group 1 and 2 previously participated in a study of postcholecystectomy pain.
  Patients in group 3 are patients scheduled for elective surgery in spinal anesthesia at the participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Spinal interleukine levels | 12 months
  12 months after surgery

SECONDARY OUTCOMES:
Blood interleukine levels | 12 Months
spinal enzyme levels | 12 months
  12 months after surgery
Blood enzyme levels | 12 months
  12 months after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense
  - Lillebælt Hospital, Vejle